CLINICAL TRIAL: NCT00868465
Title: Treatment Efficacy and Malaria TRANSmission After Artemisinin Combination Therapy (TRANSACT)
Acronym: TRANSACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); European Union (Other)
Responsible Party: Teun Bousema, Kilimanjaro Christian Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRANSACT09
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2009-04

CONDITIONS: Uncomplicated Malaria
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Artemether-lumefantrine; currently the first line treatment in Tanzania
  Interventions: Drug: Artemether-Lumefantrine
- 2 (Experimental): Dihydroartemisinin-piperaquine, alternative ACT
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Artemether-Lumefantrine — Treatment with artemether-lumefantrine (AL; Coartem; Novartis Pharma), administered as half a tablet (20 mg of artemether and 120 mg of lumefantrine) per 5 kg of body weight in a 6-dose regimen (at enrolment and 8, 20, 32, 44, and 56 h [+/-90 min] after the initiation of treatment). AL is currently the first line treatment in Tanzania
  Other Names: Coartem; Riamet
  Arms: 1
Drug: Dihydroartemisinin-piperaquine — Dihydroartemisinin-piperaquine (DP; Artekin; Duocotexin, Holley Pharm, 40 mg dihydroartemisinin/320 mg piperaquine tablets), with a dihydroartemisinin dose of 2.5 mg per kilogram and a piperaquine phosphate dose of 20 mg per kilogram daily for 3 days. DH is registered in Tanzania as Artekin and has been tested extensively in Asia and recently in clinical trials in Uganda and Rwanda
  Other Names: Artekin
  Arms: 2

SUMMARY:
Artemisinin combination therapy (ACT) with artemether lumefantrine (AL) is currently the first line treatment policy in Tanzania. AL is an efficacious drug that also has the capacity to reduce malaria transmission to mosquitoes. Nevertheless, there is concern about the development of parasite resistance against AL and there have been very few clinical trials that compared different ACT regimens. A recent clinical trial shows that the combination of dihydroartemisinin-piperaquine (DP) may be more efficacious than AL and may have a more pronounced beneficial effect on post-treatment malaria transmission. Screening for molecular markers that are related to parasite susceptibility to ACT drugs and to post-ACT treatment malaria transmission can assist in preventing the development and spread of ACT resistance.

In the current study, the investigators compared AL and DP for the treatment of uncomplicated malaria. The investigators endpoints are

* clinical efficacy
* post-treatment gametocytaemia by molecular techniques
* post-treatment malaria transmission.

DETAILED DESCRIPTION:
2.1 MALARIA AND ITS TRANSMISSION TO MOSQUITOES Malaria is the most important parasitic disease in the world. Approximately one fourth of the world population is at risk of contracting the disease, and every year more than 2 million people, mainly young children in sub-Sahara Africa, die of malaria. Malaria is caused by single-cell (protozoan) parasites of the genus Plasmodium. Four species can cause human disease: P. falciparum, P. vivax, P. ovale and P. malariae. The parasites are transmitted between humans by the bite of an infected female mosquito (Anopheles). Inside the human body, the malaria parasites multiply rapidly in the liver cells. After approximately six days, parasites leave this organ and subsequently infect red blood cells (erythrocytes). A next wave of Plasmodium replication takes place in the erythrocytes, then the red blood cell bursts, followed by infection of new red blood cells by the parasites. Since this part of the malaria life cycle involves asexual replication, parasites in this phase are referred to as asexual parasites. A small fraction of these asexual parasites develop into sexual stage parasites (gametocytes). Asexual parasites are responsible for malaria morbidity and mortality, while gametocytes ensure transmission of the parasite from humans to mosquitoes. Malaria transmission takes place when mature gametocytes are ingested by mosquitoes that are taking a blood meal. Once ingested, male and female gametocytes merge to form a zygote that develops though an ookinete stage into an oocyst that can be detected on the mosquito midgut within one week after feeding. The oocyst will burst and sporozoites are released that migrate to the mosquito salivary glands. Once the salivary glands are infected with sporozoites, the mosquito is capable of infecting new human beings.

2.2 MALARIA TREATMENT WITH ARTEMISININ COMBINCATION THERAPY (ACT) Accurate diagnosis followed by prompt and efficacious treatment is the backbone of any malaria control programme. However, malaria treatment has been facing huge challenges in recent years. A number of affordable antimalarial drugs have been used to cure malaria since the 1940s: these include chloroquine (CQ), sulphadoxine-pyrimethamine (SP; Fansidar®), mefloquine, amodiaquine (AQ) and quinine. The emergence and spread of resistance to these commonly-used drugs has been largely responsible for the worsening of the malaria situation observed in the past few years.

Across the African continent, guidelines have recently been changed. The World Health Organization (WHO) recommends for falciparum malaria the use of combination therapies, preferably those containing artemisinin derivatives (ACTs - artemisinin-based combination therapies). Artemisinin derivatives, e.g. artesunate, artemether and dihydroartemisinin, being extremely potent antimalarial agents are the ideal partners in combinations with other antimalarials. ACTs have three demonstrable advantages over conventional therapy, i) they are efficacious in treating malaria patients, ii) substantially reduce post-treatment gametocyte carriaga and iii) "protect" the partner drug from selecting resistant parasites.

In Tanzania, both CQ and SP have lost clinical efficacy. CQ was replaced by SP in 2001 and in the year 2006, SP was officially replaced by Artemether-Lumefantrine (AL: Coartem®). The policy change to the artemisinin-based drug AL is in line with the WHO recommendations to shift to ACT as first line antimalarial treatment.

2.3 RESISTANT PARASITES, MALARIA TRANSMISSION AND ACT Parasite resistance against SP has a genetic background in mutations in the parasite dihydrofolate reductase (dhfr) and dihydropteroate synthetase (dhps) genes. Single nucleotide polymorphisms (SNPs) in these genes are associated with clinical treatment failure. There is now also accumulating evidence that these mutant parasite strains also have a transmission advantage compared to wildtype parasites. Gametocyte carriage is higher for parasite with mutations in the dhfr and dhps genes, even if parasites are successfully cleared due to a longer parasite clearance time. Importantly, these mutant parasites are also more infectious to mosquitoes. These are worrying findings that may explain the rapid spread of parasite resistance in the population. The findings also indicate that gametocytes may be used as an early warning system to indicate the development of parasite resistance: parasite strains that produce most gametocytes are likely to have a reduced susceptibility to the drug.

So far, ACT has proved to be an efficient tool to reduce the transmission of malaria to mosquitoes. Compared to monotherapy with SP, ACT reduces post-treatment gametocyte prevalence and density. This translates in a reduction in post-treatment malaria transmission. Compared to monotherapy, fewer individuals are infectious to mosquitoes after ACT treatment and the average number of infected mosquitoes and the oocyst burden in mosquitoes is reduced. Importantly, ACT does not completely prevent malaria transmission but may counteract the transmission of mutant parasite strains.

2.4 ACT RESISTANCE There is a genuine fear that resistance against ACTs may develop. Although there is no direct evidence of full-blown clinical treatment failure of artemisinin derivatives, there are some worrying findings suggesting a reduced susceptibility of parasite isolates for ACTs. An increased resistance of parasite isolates to different artemisinin derivatives was observed in vitro for P. falciparum field isolates from Cambodia, French Guiana, and Senegal. This resistance was associated with SNPs at codon S769N of the ATPase6 locus of P. falciparum. In addition, the lumefantrine component of AL may exert a selective pressure for parasites with a mutation in the parasite multi-drug resistance 1 gene (Pfmdr1). In general, there is fear that there may be a selection for the artemisinin partner drugs. Although ACTs are clearly giving hopeful results, it is not yet evident which combination of drugs provides the best results, especially in the light of possible artemisinin resistance18. Recently, the combination of dihydroartemisinin-piperaquine (DP) was found to be superior to AL in reducing the risk of recurrent parasitaemia and post-treatment gametocytaemia.

Based on the finding that SP resistant parasite strains exhibit a higher gametocyte production under drug pressure, we hypothesize that gametocytaemia after treatment can be used to screen for parasites that are most likely to have a reduced susceptibility to ACT.

2. JUSTIFICATION Studies on the development of resistance to ACT and the spread of ACT resistant parasite strains in the population are extremely relevant from a public health perspective. If resistance against artemether-lumefantrine or other ACTs develops, there will be no alternative drug available for first-line treatment. The identification of predictive markers for ACT resistance will be of great value for the protection of ACT. Studies on malaria transmission after ACT are of great importance in identifying those mutations that may eventually cause ACT resistance.

The current study determines the efficacy of two different ACTs with a specific focus on detecting markers for resistance or reduced susceptibility of parasites to ACTs and the transmission potential of mutant parasites.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 10 years
* Residents of research area (5 km around the clinic)
* Willingness to come for complete scheduled follow-up.
* Uncomplicated malaria with P. falciparum mono-infection
* Parasitaemia of 1000-200,000 parasites/ul
* Temperature > 37.5°C and < 39.5°C, or history of fever in previous 24 hours.
* No history of adverse reactions to AL
* Understanding of the procedures of the study by parent or guardian and willing to participate by signing informed consent forms.

Exclusion Criteria:

* General signs of severe malaria
* Haemoglobin concentration < 5g/dl
* Presence of disease other than malaria causing febrile conditions
* Mixed infection with P. malariae or other non-falciparum malaria species
* Unwilling to participate and sign informed consent forms.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the clinical efficacy of artemether-lumefantrine (AL) and dihydroartemisinin-piperaquine (DP) in the treatment of uncomplicated falciparum malaria in children living in north-western Tanzania and in western Kenya. | during 42 day follow-up

SECONDARY OUTCOMES:
To determine (sub-microscopic) gametocyte carriage after treatment with AL and DP | during 42 day follow-up
To determine malaria transmission to mosquitoes after treatment with AL or DP | day 7 after initiation treatment
To determine molecular markers that are predictive of reduced susceptibility of parasite strains for AL and DP | day 7 after initiation treatment
To determine molecular markers that are related to gametocytaemia or malaria transmission after treatment with AL and DP | during 42 day follow-up
To determine the relation between treatment success and the presence of anti-malaria antibodies | during 42 day follow-up
To explore the role of cellular oxidative stress in treatment with AL and DP | during 42 day follow-up
To determine the relation between transmission to mosquitoes and the presence of anti-malaria antibodies | day 7 after initiation treatment

CONTACTS AND LOCATIONS:
Locations (2):
- International Centre for Insect Physiology and Ecology - St. Judes Clinic, Mbita, Suba District, Kenya
- Kilimanjaro Christian Medical Centre, Magugu Field Site, Moshi, Kilimanjaro, Tanzania

REFERENCES:
- [Background] Bousema JT, Schneider P, Gouagna LC, Drakeley CJ, Tostmann A, Houben R, Githure JI, Ord R, Sutherland CJ, Omar SA, Sauerwein RW. Moderate effect of artemisinin-based combination therapy on transmission of Plasmodium falciparum. J Infect Dis. 2006 Apr 15;193(8):1151-9. doi: 10.1086/503051. Epub 2006 Mar 15. PMID 16544256
- [Background] Hallett RL, Sutherland CJ, Alexander N, Ord R, Jawara M, Drakeley CJ, Pinder M, Walraven G, Targett GA, Alloueche A. Combination therapy counteracts the enhanced transmission of drug-resistant malaria parasites to mosquitoes. Antimicrob Agents Chemother. 2004 Oct;48(10):3940-3. doi: 10.1128/AAC.48.10.3940-3943.2004. PMID 15388456
- [Derived] Muwanguzi J, Henriques G, Sawa P, Bousema T, Sutherland CJ, Beshir KB. Lack of K13 mutations in Plasmodium falciparum persisting after artemisinin combination therapy treatment of Kenyan children. Malar J. 2016 Jan 22;15:36. doi: 10.1186/s12936-016-1095-y. PMID 26801909
- [Derived] Sawa P, Shekalaghe SA, Drakeley CJ, Sutherland CJ, Mweresa CK, Baidjoe AY, Manjurano A, Kavishe RA, Beshir KB, Yussuf RU, Omar SA, Hermsen CC, Okell L, Schallig HD, Sauerwein RW, Hallett RL, Bousema T. Malaria transmission after artemether-lumefantrine and dihydroartemisinin-piperaquine: a randomized trial. J Infect Dis. 2013 Jun 1;207(11):1637-45. doi: 10.1093/infdis/jit077. Epub 2013 Mar 6. PMID 23468056